CLINICAL TRIAL: NCT05236764
Title: T-Cell Receptor Alpha Beta+/CD19+ Depletion in Haploidentical Allogeneic Hematopoietic Cell Transplantation (Allo-HCT) for Adult and Pediatric Patients With Hematological Malignancies and Non-malignant Disorders
Brief Title: Haploidentical Hematopoietic Cell Transplantation Using TCR Alpha/Beta and CD19 Depletion
Acronym: HAPLOTAB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Erin Morales, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-50045 HAPLOTAB
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Myelodysplastic Syndromes; Chronic Myeloid Leukemia; Hemophagocytic Lymphohistiocytoses; Primary Immunodeficiency Diseases; Hemoglobinopathies; Severe Aplastic Anemia; Cytopenia; Bone Marrow Failure Syndrome; Severe Chronic Active Epstein-Barr Virus Infection
Keywords: Stem Cell Transplant; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Non-Hodgkins Lymphoma; Chronic Myeloid Leukemia; Hemophagocytic Lymphohistiocytoses; Primary Immunodeficiency Diseases; Hemoglobinopathies; Severe Aplastic Anemia; Congenital/hereditary cytopenias including Fanconi Anemia; Bone Marrow Failure Syndrome; Severe Chronic active Epstein-Barr Virus Infections
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphohistiocytosis, Hemophagocytic; Primary Immunodeficiency Diseases; Hemoglobinopathies; Anemia, Aplastic; Cytopenia; Bone Marrow Failure Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Alpha beta+ T cell depleted CD34+ stem cells (Experimental): The patient will be receiving a donor stem cell transplant with a preceding conditioning regimen (chemotherapy with, or without, radiation). The investigators will be specially treating the donor's blood cells used for the stem cell transplant.
  Interventions: Device: CliniMACS

INTERVENTIONS:
Device: CliniMACS — Peripheral blood stem cells from closely matched unrelated donors will be processed using the CliniMACS device to remove TCRalpha/beta (alpha beta+) T cells and B cells, in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique

SUMMARY:
Patients with medical conditions requiring allogeneic hematopoietic cell transplantation (allo-HCT) are at risk of developing a condition called graft versus host disease (GvHD) which carries a high morbidity and mortality. This is a phase I/II study that will test the safety and efficacy of hematopoietic cell transplantation (HCT) with ex-vivo T cell receptor Alpha/Beta+ and CD19 depletion to treat patients' underlying condition. This process is expected to substantially decrease the risk of GvHD thus allowing for the elimination of immunosuppressive therapy post-transplant. The study will use blood stem/progenitor cells collected from the peripheral blood of parent or other half-matched (haploidentical) family member donor. The procedure will be performed using CliniMACS® TCRα/β-Biotin System which is considered investigational.

DETAILED DESCRIPTION:
This is a phase I/II study of haploidentical HCT (HHCT) with ex vivo TCRαβ+ and CD19+ depletion using the CliniMACS device in patients with hematological malignancies and non-malignant disorders. HHCT will be performed according to current standards of care at the Center for Cell and Gene Therapy (CAGT) within Texas Children's Hospital (TCH) and Houston Methodist Hospital (HMH), including the use of a standard chemotherapy conditioning regimens, supportive care and standard follow-up laboratory assessments. The study will determine efficacy of this strategy in terms of engraftment, and safety in terms of rates of acute and chronic graft versus Host Disease (GvHD), one-year overall survival (OS) and transplant-related mortality (TRM).

The peripheral blood hematopoietic cell product will undergo negative selection of TCR αβ following the standardized protocol in the user's manual for the CliniMACS (Miltenyi Biotech, Germany). TCR αβ+ T-cells are labeled by CliniMACS TCR αβ-Biotin (murine anti-TCR αβ monoclonal antibodies conjugated to biotin) which allows the TCR αβ+ T-cells to be magnetically labeled with CliniMACS Anti-Biotin Microbeads (murine anti-biotin monoclonal antibodies conjugated to superparamagnetic iron dextran particles) for depletion. The CD19+ B cells are labeled by CliniMACS CD19 microbeads which allows the CD19+ B cells to be magnetically labeled for depletion. All unlabeled cells are selected as target cells which should contain a minimum amount of TCR αβ+ and CD19+ cells. The microbeads used for labeling are approximately 50 nanometers in diameter and do not require removal prior to patient infusion.

In January 2014, the U.S. Food and Drug Administration (FDA) has approved the Miltenyi Biotec's CliniMACS CD34 Reagent System as a Humanitarian Use Device for the prevention of GvHD in patients with acute myeloid leukemia (AML) in first complete remission undergoing allo-HCT from HLA-matched related donor.

ELIGIBILITY:
Inclusion Criteria:

1. Lack of suitable conventional donor (10/10 HLA matched related or unrelated donor) or presence of rapidly progressive disease not permitting time to identify an HLA-matched unrelated donor. This does not include cord blood unit (CBU) availability.
2. Lansky/Karnofsky score > 50
3. Signed written informed consent
4. Diagnosis of one of the following:

   1. Patient with life threatening hematological malignancy including "high-risk" ALL in first complete remission (CR1); ALL in second or subsequent remission (greater than or equal to CR2); high-risk AML in CR1; AML in second or subsequent CR; myelodysplastic syndromes (MDS); non-Hodgkin's lymphomas (NHL) in second or subsequent remission (greater than or equal to CR2); CML
   2. Hemophagocytic Lymphohistiocytosis (HLH) including familial HLH, relapsed HLH or central nervous system (CNS) HLH
   3. Primary Immunodeficiency Disorders (PID)
   4. Hemoglobinopathies including thalassemia or sickle cell disease (SCD)
   5. Severe aplastic anemia (SAA) not responding to immune suppressive therapy
   6. Congenital/hereditary cytopenias including Fanconi anemia (FA) without malignant clonal evolution (MDA, AML)
   7. Other inherited bone marrow failure syndromes (IBMFS)
   8. Sever chronic active Epstein Barr virus infection (SCAEBV) with predilection for T-or NK-cell malignancy

NOTE: 'High risk' ALL or AML refers to those acute leukemias identified by the presence of specific biologic features, which predict high likelihood of failure to conventional chemotherapy. As biologic features of high-risk disease evolve with improvement of conventional chemotherapy, it is not practical to define this indication with any further specificity. Therefore, high risk AML/ALL will be determined by the primary physician.

Exclusion Criteria:

1. Life expectancy of less than or equal to 6 weeks
2. Greater than grade II acute graft versus host disease (GVHD) or chronic extensive GVHD due to a previous allograft at the time of inclusion
3. Subject receiving an immunosuppressive treatment for GVHD treatment due to a previous allograft at the time of inclusion
4. Symptomatic cardiac disease or left ventricular shortening fraction less than 25% or ejection fraction < 40%
5. Severe renal disease, with creatinine clearance < 40cc/1.73m2
6. Pre-existing severe restrictive pulmonary disease, FVC < 40% of predicted
7. Severe Hepatic Disease with ALT/AST ≥ x 2.5 upper limit of normal or bilirubin level ≥ x 1.5 upper limit of normal
8. Serious concurrent uncontrolled medical disorder or mental illness
9. Pregnant or breastfeeding female subject
10. Current active infectious disease including viral and fungal diseases at the time of enrollment; that on evaluation of PI precludes ablative chemotherapy or successful transplantation
11. Active HIV infection
12. Severe personality disorder or mental illness that would preclude compliance with the study

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2026-05-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Morales, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha beta+ T cell depleted CD34+ stem cells
Started | 3
Completed | 0
Not Completed | 3
Not completed — In follow up (ongoing) | 1
Not completed — Taken off study - secondary graft failure | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alpha Beta+ T Cell Depleted CD34+ Stem Cells
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Neutrophil Engraftment and Platelet Engraftment
Description: Cumulative incidence of neutrophil and platelet engraftment (composite measure) will be reported as rate and its associated 95% confidence interval. Competing risks methods will be utilized, with graft failure and death considered as competing risks.
  Neutrophil engraftment is defined as the first of 3 consecutive days with a peripheral blood absolute neutrophil count of ≥ 0.5x10^9/L
  Platelet engraftment is defined as the first day with platelet count of ≥ 20 x10^9/L without transfusion support for 7 consecutive days
Time Frame: 42 days post-HCT
Population: All patients who received transplant were included in analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Alpha beta+ T cell depleted CD34+ stem cells
Number analyzed (Participants) | 3
Percentage of participants | 66.7 [0.2 to 97.3]

2. Primary Outcome: Cumulative Incidence of Grade III or Higher Acute GVHD
Description: Cumulative incidence of grade III or higher acute GVHD among patients who achieve engraftment will be reported as rate and its associated 95% confidence interval. Competing risks methods will be utilized, with death considered the competing risk.
Time Frame: 100 days post-HCT
Population: All patients who received transplant and did not encounter graft failure are included in analysis. Patients who had graft failure were not evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Alpha beta+ T cell depleted CD34+ stem cells
Number analyzed (Participants) | 2
Percentage of participants | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Cumulative Incidence of Transplant-related Mortality (TRM)
Description: Cumulative incidence of transplant related mortality will be reported as rate and its associated 95% confidence interval.
  TRM is defined as death due to any transplantation-related cause, other than disease
Time Frame: 100 days and 365 days post-HCT
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the day of transplant to death
Time Frame: Up to one year post-HCT
Reporting Status: Not Posted

5. Secondary Outcome: Cumulative Incidence of Chronic Graft Versus Host Disease
Description: Cumulative incidence of chronic GVHD among patients who achieve engraftment will be reported as rate of chronic GvHD and its associated 95% confidence interval.
Time Frame: Up to two years post HCT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 until 30-days post-transplant for adverse events, and until 100-days post-transplant for serious adverse events.
Arm/Group | Alpha beta+ T cell depleted CD34+ stem cells
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha beta+ T cell depleted CD34+ stem cells (N=3)
Fever (General disorders and administration site conditions) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Viremia (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha beta+ T cell depleted CD34+ stem cells (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT05236764/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT05236764/ICF_002.pdf